CLINICAL TRIAL: NCT01524952
Title: The Effect of Combined Thermal and Electrical Muscle Stimulation (cTEMS) on Cardiorespiratory Fitness and Adipose Tissue in Obese Individuals
Brief Title: The Effect of Combined Thermal and Electrical Muscle Stimulation (cTEMS) on Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009/1273
Record Dates: First submitted 2012-01-25; First posted 2012-02-02 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active (Experimental): cTEMS
  Interventions: Device: combined thermal and electrical muscle stimulation (cTEMS)

INTERVENTIONS:
Device: combined thermal and electrical muscle stimulation (cTEMS) — cTEMS in three 60-minute sessions per week for 8 weeks

SUMMARY:
Objective:

It is unclear whether prolonged electrical muscle stimulation can improve cardiorespiratory fitness and reduce body fat in obese subjects. The purpose of this study is to investigate the effect of prolonged combined thermal and electrical muscle stimulation (cTEMS) on peak oxygen consumption (VO2 peak) and body composition. We will also investigate the biochemical effects and the resultant lipolysis-related gene expression changes in adipocytes.

Methods:Eleven obese (BMI≥30) individuals will receive cTEMS in three 60-minute sessions per week for 8 weeks. Activity levels and dietary habits will be kept unchanged and controlled with an accelerometer and nutritional questionnaire. Before and after the stimulation period, functional capacity are assessed by VO2 peak, and body composition was assessed by dual-energy X-ray absorptiometry and bioelectrical impedance analyses. Lipolytic activity will be determined in abdominal adipose tissue by 24 hours of microdialysis on a sedentary day, and adipose tissue biopsies will be taken for the gene expression analysis.

ELIGIBILITY:
Inclusion Criteria:

* Obese (Body mass index; BMI ≥ 30 kg/m2),
* sedentary subjects (< 20 minutes of exercise < 3 days per week).
* Other inclusion criteria were age between 30 and 70 years and
* the ability to undergo exercise testing.

Exclusion Criteria:

* Pacemaker or implanted defibrillator,
* regular medication,
* cardiovascular disease,
* pulmonary disease,
* extensive dermatological disease or other primary diseases;
* pregnant women;
* and individuals who abuse alcohol or drugs were excluded from the study

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-12; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Oxygen uptake | Baseline and after 10 weeks

SECONDARY OUTCOMES:
Lipolytic activity | Baseline and after 10 weeks
  Lipolytic activity in adipose tissue measured by microdialysis
Gene expression in adipose tissue | Baseline and after 10 weeks
Body composition | Baseline and after 10 weeks
  Body composition by DEXA

CONTACTS AND LOCATIONS:
Overall Officials: Jan Erik Nordrehaug, PhD, Study Chair — University of Bergen
Locations (1):
- Haukeland University Hospital, Bergen, Norway